CLINICAL TRIAL: NCT02826421
Title: Clinical Investigation of Corneal Incision Size After IOL Implantation With Preloaded Delivery Devices and a Manual Delivery Device
Brief Title: Clinical Investigation of Corneal Incision Size After Intraocular Lens (IOL) Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILN296-P001
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-07

CONDITIONS: Cataracts
Keywords: Intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- UltraSert Preloaded Delivery System (Experimental): Preloaded IOL delivered via a 2.2 mm clear corneal incision during cataract surgery
  Interventions: Device: UltraSert Preloaded Delivery System
- iTec Preloaded Delivery System (Active Comparator): Preloaded IOL delivered via a 2.2 mm clear corneal incision during cataract surgery
  Interventions: Device: iTec Preloaded Delivery System
- iSert Preloaded Delivery System (Active Comparator): Preloaded IOL delivered via a 2.2 mm clear corneal incision during cataract surgery
  Interventions: Device: iSert Preloaded Delivery System
- Monarch III D Manual IOL Delivery System (Active Comparator): Manually loaded IOL delivered via a 2.4 mm clear corneal incision during cataract surgery
  Interventions: Device: Monarch III D Manual IOL Delivery System

INTERVENTIONS:
Device: UltraSert Preloaded Delivery System — Includes AcrySof IQ monofocal posterior chamber IOL Model AU00T0, intended for long term use over the lifetime of the subject
  Arms: UltraSert Preloaded Delivery System
Device: iTec Preloaded Delivery System — Includes TECNIS 1-piece monofocal IOL, intended for long term use over the lifetime of the subject
  Arms: iTec Preloaded Delivery System
Device: iSert Preloaded Delivery System — Includes Model 251 or Model 250 posterior chamber IOL, as selected by the Investigator, intended for long term use over the lifetime of the subject
  Arms: iSert Preloaded Delivery System
Device: Monarch III D Manual IOL Delivery System — Includes AcrySof IQ monofocal IOL posterior chamber IOL Model SN60WF, intended for long term use over the lifetime of the subject
  Arms: Monarch III D Manual IOL Delivery System

SUMMARY:
The purpose of this study is to compare corneal incision size after IOL implantation with the use of one of four IOL delivery systems (three preloaded IOL delivery systems and one manually loaded IOL delivery system).

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and sign a statement of informed consent;
* Willing and able to complete all required postoperative visits;
* Cataract;
* Planned cataract removal by phacoemulsification;
* Calculated lens power from 18.0 through 27.0 D inclusive;
* Preoperative astigmatism <1.0D;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Systemic disease that affects the cornea;
* Any inflammation or edema of the cornea;
* Previous or planned refractive or corneal surgery during the subject's participation in the study;
* Previous corneal transplant;
* Previous retinal detachment;
* Pregnancy or lactation, current or planned, during the course of the study;
* Current participation in another investigational drug or device study that may confound the results of this investigation;
* Any condition observed before or during surgery that in the surgeon's medical opinion may affect the success of the cataract surgery;
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, GCRA, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 study centers located in Spain and 2 study centers located in France.
Pre-assignment Details: Of the 114 enrolled, 2 subjects did not meet inclusion/exclusion criteria, and 3 subjects were excluded prior to randomization for "other" reasons (ie, the maximum number of randomized subjects was reached). This reporting group includes all randomized subjects (109).
Groups:
- UltraSert; iTec; iSert: Preloaded IOL delivered via a 2.2 mm clear corneal incision during cataract surgery
- Monarch III D: Manually loaded IOL delivered via a 2.4 mm clear corneal incision during cataract surgery
Period: Overall Study
Arm/Group | UltraSert | iTec | iSert | Monarch III D
Started | 22 | 29 | 28 | 30
Treated | 19 | 26 | 26 | 28
Completed | 19 | 26 | 26 | 28
Not Completed | 3 | 3 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 1 | 1
Not completed — Reason not given | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects whose cataract surgery procedure was completed (Full Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | UltraSert | iTec | iSert | Monarch III D | Total
Number analyzed (Participants) | 19 | 26 | 26 | 28 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (8.71) | 70.7 (8.31) | 73.0 (7.27) | 72.5 (7.10) | 71.9 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 14 | 17 | 58
  Male | 5 | 13 | 12 | 11 | 41

OUTCOME MEASURES:

1. Primary Outcome: Mean Corneal Incision Size After IOL Implantation (UltraSert, iTec, and iSert)
Description: Post-IOL implantation corneal incision size was measured directly after IOL implantation and reported in millimeters (mm). Minimizing enlargement of incision size during cataract surgery results in less postoperative inflammation, less surgically-induced astigmatism, and more rapid visual and wound rehabilitation. This endpoint was prespecified for the UltraSert, iTec, and iSert preloaded delivery systems. Only one eye (study eye) contributed to the analysis.
Time Frame: Day 0, operative day
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: mm
Arm/Group | UltraSert | iTec | iSert
Number analyzed (Participants) | 19 | 26 | 26
mm | 2.35 (0.019) | 2.47 (0.016) | 2.54 (0.019)

2. Secondary Outcome: Mean Corneal Incision Size After IOL Implantation (UltraSert and Monarch III D)
Description: Post-IOL implantation corneal incision size was measured directly after IOL implantation and reported in millimeters (mm). Minimizing enlargement of incision size during cataract surgery results in less postoperative inflammation, less surgically-induced astigmatism, and more rapid visual and wound rehabilitation. This endpoint was prespecified for the UltraSert preloaded delivery system and the Monarch III D delivery system. Only one eye (study eye) contributed to the analysis.
Time Frame: Day 0, operative day
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: mm
Arm/Group | UltraSert | Monarch III D
Number analyzed (Participants) | 19 | 28
mm | 2.35 (0.019) | 2.49 (0.011)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 31 days). AEs are reported as pretreatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the medical device. Ocular adverse events are presented for both study eye and non-study eye combined.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to initiation of study treatment
- UltraSert: All subjects treated with UltraSert
- iTec: All subjects treated with iTec
- iSert: All subjects treated with iSert
- Monarch III D: All subjects treated with Monarch III D
Arm/Group | Pretreatment | UltraSert | iTec | iSert | Monarch III D
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/19 | 0/26 | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/114 | 0/19 | 1/26 | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 0/114 | 0/19 | 0/26 | 0/26 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=114) | UltraSert (N=19) | iTec (N=26) | iSert (N=26) | Monarch III D (N=28)
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Surgical procedure repeated (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.